CLINICAL TRIAL: NCT04397848
Title: Hearing and Supporting the Healthcare Workers: Mental Health Outcomes in Healthcare Workers During COVID-19
Brief Title: Mental Health Outcomes in Healthcare Workers During COVID-19
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: William Osler Health System (Other); University of Toronto (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Rima Styra, Dr. Rima Styra, MD,MEd, FRCPC, ABPN, University Health Network, Toronto
Other Study IDs: 3189
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Mental Health Wellness 1; PTSD; Anxiety; Stress; Depression; COVID-19; Healthcare Workers
Keywords: Healthcare Workers; COVID-19; Mental Health Outcomes
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An online survey will be sent to healthcare workers (HCWs) in acute care hospitals to explore a variety of risk factors for negative psychological outcomes and levels of anxiety, depression and post-traumatic stress symptoms using validated scales. It is important to understand the sources of negative psychological impact on HCWs during this COVID-19 pandemic before hospitals and organizations can address and develop support programs to mitigate the stresses experienced by healthcare workers. Addressing and supporting the needs of our HCWs will be paramount in this COVID-19 pandemic and future outbreaks.

DETAILED DESCRIPTION:
Previous work conducted by our group during the 2003 SARS outbreak demonstrated symptoms of post-traumatic stress disorder (PTSD) and depression in healthcare workers (HCWs) working in high-risk areas. Similar reports are emerging with regards to HCWs during COVID-19 which may affect staff mental health outcomes which may have effects on staff absenteeism and retention.

The study is a cross-sectional, multi-centered, hospital-based online survey conducted at several Toronto hospitals. Participants will be recruited to participate in the voluntary study via an internal e-mail that will contain a short description of the study and a link to the online survey. The survey will take approximately 25 minutes to complete. The study group will include HCW s from high-risk units (Emergency, ICU, and COVID-19 units) with a comparison group of HCWs who are not directly involved in the assessment or management of patients with COVID-19.

This study will evaluate the psychological impact of the COVID-19 pandemic on HCW's and identify risk factors that may place HCWs at greater risk for negative psychological outcomes. The survey will gather information such as s basic, non-identifying demographic information, hospital and unit of work, quarantine and isolation, work with patients diagnosed with COVID-19, loss of loved ones to COVID-19, understanding of the reasons for PPE/ infection control directives, perceptions of risk to self and family, sources of support. As well, Toronto is in the unique situation of having been at the centre of the 2003 Canadian SARS outbreak and presently experiencing the impact of the COVID-19. The investigators propose that COVID-19 might have a differential impact on the psychological wellbeing of current HCWs depending on whether they practiced during SARS. Our survey will explore the differences of the psychological impact of the COVID-19 pandemic on healthcare workers who lived through the SARS outbreak and those who did not. The following validated scales are embedded in the survey to evaluate the psychological impact of the COVID pandemic: Impact of Event Scale-Revised (IES-R), Generalized Anxiety Disorder -7 (GAD-7) , and Patient Health Questionnaire (PHQ-9). Open-ended questions will also provide respondents the opportunity to relate aspects of working during the COVID-19 pandemic that are most difficult and to provide additional comments on their unique experiences.

ELIGIBILITY:
Inclusion Criteria:

HCW currently working at Toronto based hospitals: University Health Network (UHN), Sunnybrook Health Sciences and William Osler Health System.

Exclusion Criteria: Not a healthcare worker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group will include all HCWs working within the hospital system. This will include HCWs from high-risk units such as Emergency, ICU, and COVID-19 units as well as HCWs who are not directly involved in the assessment or management of patients with COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 3852 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Impact of Event Scale - Revised (IES-R) | Two weeks
  Scale to evaluate Post-traumatic Stress Disorder symptoms
General Anxiety Disorder (GAD-7) | Two weeks
  Scale to evaluate anxiety symptoms
Patient Health Questionnaire (PHQ-9) | Two weeks
  Scale to evaluate depressive symptoms

SECONDARY OUTCOMES:
Qualitative Data | Two weeks
  Qualitative data will be coded and analyzed to show emerging themes.

CONTACTS AND LOCATIONS:
Overall Officials: Rima Styra, MD, MEd, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada